CLINICAL TRIAL: NCT01369732
Title: Prevention of Acute Kidney Injury by Erythropoietin in Patients Undergoing Thoracic Aorta Surgery With Hypothermic Cardiac Arrest
Brief Title: Prevention of Acute Kidney Injury by Erythropoietin in Thoracic Aorta Surgery With Hypothermic Cardiac Arrest
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3-2011-0086
Record Dates: First submitted 2011-06-03; First posted 2011-06-09 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-07

CONDITIONS: Dissection of Thoracic Aorta
MeSH Terms: conditions — Dissection, Thoracic Aorta | interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline group (Placebo Comparator): We administrate the saline single bolus (5ml, intravenously) 30 min before the commencement of ischemia.
  Interventions: Drug: saline
- erythropoietin group (Experimental): We administrate the erythropoietin single bolus (500 IU/kg intravenously) 30 min before the commencement of ischemia.
  Interventions: Drug: recombinant human erythropoietin

INTERVENTIONS:
Drug: recombinant human erythropoietin — We administrate the erythropoietin single bolus (500 IU/kg intravenously) 30 min before the commencement of ischemia.
  Other Names: epocaine
  Arms: erythropoietin group
Drug: saline — We administrate the saline single bolus (5ml intravenously) 30 min before the commencement of ischemia.
  Other Names: normal saline
  Arms: Saline group

SUMMARY:
During thoracic aortic surgery, hypothermic cardiac arrest causes aortic ischemia and reperfusion (IR) periods, respectively. Aortic ischemia results in an ischemic insult to the lower extremities and successive reperfusion results in injury to remote organs, including kidneys. So, there has been considerable interest in the development of therapeutic strategies aimed at attenuating IR injury. One such group of agents that are attracting interest due to their potential protective effects on vascular endothelium is the erythropoietin.

However, the effect of erythropoietin on renal injury induced by aortic IR in humane has not been fully clarified. Therefore, the purpose of this study is to determine whether the prophylactic administration of erythropoietin reduce the incidence of acute kidney injury (AKI) in patients undergoing thoracic aorta surgery with hypothermic cardiac arrest. The investigators administrate the erythropoietin single bolus (500 IU/kg intravenously) 30 min before the commencement of ischemia. The differences between the control and study groups are observed by clinical indicators such as serum creatinine, TNF-α, NGAL.

ELIGIBILITY:
Inclusion Criteria:

1. Adults above age of 20
2. Undergoing Thoracic Aorta Surgery with Hypothermic Cardiac Arrest

Exclusion Criteria:

1. pregnancy or lactation
2. cerebrovascular thrombosis 3. past history of pulmonary embolism or thrombosis
3. past history of thoracic aortic surgery
4. malignancy 5. preoperative acute kidney injury
5. chronic renal replacement therapy
6. allergy or hypersensitivity to erythropoetin
7. history of erythropoetin treatment
8. death during or one day after surgery
9. no consent
10. reoperation within seven days of the first surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yon Hee Shim, Study Director — Yonsei University
Locations (1):
- Gangnam severance hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at the university hospital between May 2011 and January 2013.
Pre-assignment Details: Six patients were dropped out regarding wrong dose-count of erythropoietin (n = 1), death within 24 hours after surgery (n = 2), and screening failure due to chronic kidney disease (n = 3).
Period: Overall Study
Arm/Group | Saline Group | Erythropoietin Group
Started | 33 | 33
Completed | 29 | 31
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline Group | Erythropoietin Group | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 20 | 37
  >=65 years | 16 | 13 | 29
Age Continuous [Mean (Standard Deviation); unit: years] | 65 (12) | 61 (13) | 63 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 20 | 31
  Male | 22 | 13 | 35
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Acute Kidney Injury Based on RIFLE Criteria
Description: Serum creatinine, GFR, urine output will be measured at 6:00 AM everyday up to 7 days after surgery.
Time Frame: upto 7 days after surgery
Reporting Status: Not Posted

2. Secondary Outcome: Mortality
Description: Participants will be followed for the mortality, an expected average of 1 month after surgery.
Time Frame: upto 1 month after surgery
Reporting Status: Not Posted

3. Secondary Outcome: the Duration of Mechanical Ventilation
Description: Participants will be followed for the duration of mechanical ventilation, an expected average of 2 weeks after surgery.
Time Frame: upto 2 weeks after surgery
Reporting Status: Not Posted

4. Secondary Outcome: the Duration of ICU Stay
Description: Participants will be followed for the duration of ICU stay, an expected average of 2 weeks after surgery.
Time Frame: upto 2 weeks after surgery
Reporting Status: Not Posted

5. Secondary Outcome: the Duration of Hospital Stay
Description: Participants will be followed for the duration of hospital stay, an expected average of 1 month after surgery.
Time Frame: upto 1 month after surgery
Reporting Status: Not Posted

6. Primary Outcome: Incidence of Acute Kidney Injury Based on RIFLE Criteria
Time Frame: upto 7 days after surgery
Measure: Number; unit: participants
Arm/Group | Saline Group | Erythropoietin Group
Number analyzed (Participants) | 29 | 31
participants | 18 | 18

ADVERSE EVENTS:
Arm/Group | Saline Group | Erythropoietin Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No